CLINICAL TRIAL: NCT05418374
Title: Effects of Continuous Versus Single Dose Spinal Anesthesia in Octagenerians Undergoing Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU 54/2022
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Octagenerian Population Undergoing Hip Surgeries
Keywords: Octagenerians; Hip surgery; Spinal anesthesia; Continuous spinal anesthesia; Visual Analogue Scale

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 18G epidural needle will be inserted intrathecally at the level of L4-L5. After insertion of the Tuohy needle, the subarachnoid space is found and the bevel is directed downward, and the spinal catheter is passed 2-3 cm into the subarachnoid space. After confirmation of aspiration cerebral spinal fluid through the catheter, an initial dose 2.5 mg (0.5 ml) of plain bupivacaine 0.5%(manufactured by sunny medical ) will be injected.
  Interventions: Procedure: Continous Spinal Anestheisa
- Control group (No Intervention): traditional spinal anesthesia will be done with a 25G pencil point spinal needle at the level of L4-L5 with injection of 12.5 mg (2.5ml) of bupivacaine 0.5%. By adjusting the head level, T10 sensory block will be targeted

INTERVENTIONS:
Procedure: Continous Spinal Anestheisa — Continuous spinal anesthesia (CSA) describes subarachnoid blockade maintained by local anesthetics administered through an indwelling spinal catheter. CSA provides fewer episodes of hypotension and no severe hypotension versus single dose bupivacaine also it offers the ability to titrate the dose of local anesthetics needed while maintaining hemodynamic stability.
  Arms: Group A

SUMMARY:
Continuous spinal anesthesia (CSA) is an anesthetic technique that offers several clinical advantages for anesthesia and analgesia in elderly patients. The level of sensory blockade can be titrated to the desired dermatomal level with great precision with intrathecal (IT) catheters, allowing better control of the hemodynamic consequences of sympathetic blockade associated with spinal anesthesia compared to epidural or single shot spinal techniques. Better control of hemodynamics maybe advantageous in patients with cardiac disease in whom administration of lower doses of local anesthetics is advantageous. Greater numbers of patients are presenting for surgery with aging-related pre-existing conditions, which places them at greater risk of an adverse outcome, such as cardiac or pulmonary disease or diabetes mellitus. CSA allows incremental dosing of an intrathecal local anesthetic providing fewer hemodynamic alterations. While spinal anesthesia is widely used anesthetic technique in lower limb surgery in the elderly, it induces more hemodynamic instability due to high blockage effect which largely limits the use of conventional dose of spinal anesthesia in high risk elderly patients

DETAILED DESCRIPTION:
METHODOLOGY:

Patients and Method. Type of Study: Randomized controlled clinical trial. Approval will be obtained from the research ethics committee of Faculty of Medicine; Ain Shams University and a written informed consent will be taken from each patient to participate in the study. Study Setting: Ain-shams University Hospitals, Cairo, Egypt. Study Period: 6 months from approval of medical ethics committee. Sample Size: Based on the study of continuous spinal Anestheisa by Vincent M, Olivier F, and David G, 2006 assuming a rate of hypotension attacks (20% of the baseline blood pressure) of 15% in CSA group compared to 65% in SD spinal anesthesia group, a sample of 20 patients in each group is enough to detect such METHODOLOGY: Patients and Method. Type of Study: Randomized controlled clinical trial. Approval will be obtained from the research ethics committee of Faculty of Medicine; Ain Shams University and a written informed consent will be taken from each patient to participate in the study.METHODOLOGY:

Patients and Method. Type of Study: Randomized controlled clinical trial.

Study Setting: Ain-shams University Hospitals, Cairo, Egypt. Study Period: 6 months from approval of medical ethics committee. Sample Size: Based on the study of continuous spinal Anestheisa by Vincent M, Olivier F, and David G, 2006 (3) assuming a rate of hypotension attacks (20% of the baseline blood pressure) of 15% in CSA group compared to 65% in SD spinal anesthesia group, a sample of 20 patients in each group is enough to detect such difference, at 0.05 alpha error and 80% power of the test. Study tool: Visual Analogue Scale (VAS)

Study Procedures:

Based on this data, patients will be randomly allocated into two groups with 20 patients in each group.

A. Preoperative settings:

All patients will be assessed preoperatively by careful history taking, full physical examination, and laboratory evaluation according to institutional guidelines, ECG and ECHO. A written consent will be taken after full description of the procedure. The Visual Analogue Score will be described properly to the patient before the procedure.

. Intraoperative settings: Patient will be allocated in one of the 2 study groups, Group A will receive continuous spinal anesthesia and Group B (control group) will receive traditional spinal anesthesia, All standard monitors will be placed (NIBP, pulse oximeter and electrocardiogram). All patients will receive oxygen (3 L/min) during the procedure, including the first postoperative hours. All patients will have an intravenous line (18G cannula), 500 ml Ringer will be started as a preload, airway and resuscitation equipment will be readily available. All equipment for the spinal blockade will be ready for use, and all necessary medications will be drawn up prior to positioning the patient for spinal anesthesia. Patients will receive 0.4 mg/kg propofol IV 3 min before being turned to the lateral position for lumbar puncture. The patient will be positioned in lateral position with the injured leg up. The ideal positioning consists of having the back of the patient parallel to the edge of the bed closest to the anesthesiologist, with the patient's knees flexed to the abdomen and neck flexed, the midline will be palpated. The iliac crests will be palpated, and a line is drawn between them to find the body of L4 or the L4-L5 interspace. All techniques will be done under complete aseptic condition using Betadine 5%. A small wheal of local anesthetic (lidocaine 0.5%) is injected into the skin at the planned site of insertion. In study group (A), 18G epidural needle will be inserted intrathecally at the level of L4-L5. After insertion of the Tuohy needle, the subarachnoid space is found and the bevel is directed downward, and the spinal catheter is passed 2-3 cm into the subarachnoid space. After confirmation of aspiration cerebral spinal fluid through the catheter, an initial dose 2.5 mg (0.5 ml) of plain bupivacaine 0.5%(manufactured by sunny medical ) will be injected. After assessment of systemic blood pressure and sensory level, After completion of injection the patients remained in the lateral position for 5 min and then will be returned to the supine position, increments of 2.5 mg (0.5 ml) of the same solution will be given every 15 minutes until reaching the required anesthetic level of T10. In case of failure or insufficient block, general anesthesia will be performed. In control group traditional spinal anesthesia will be done with a 25G pencil point spinal needle at the level of L4-L5 with injection of 12.5 mg (2.5ml) of bupivacaine 0.5%. By adjusting the head level, T10 sensory block will be targeted. In both groups, patients will be positioned for surgery after achieving sensory blockage of T10 level. Testing the sensory level will be done using The ice pack method: by Placing an ice on an area well away from the possible dermatome cover (eg face or forearm) and ask them to tell you how cold it feels to them then Apply the ice to an area likely to be blocked on the same side of the body and ask the patient "Does this feel the same cold as your face/arm or different?" Patients may report the ice feeling colder, warmer or the same, Apply the ice to areas above and below this point until it's clear at which level the top and the bottom of the block is and repeat the procedure on the opposite side of the body continuous close monitoring of vital data and complications of spinal anesthesia will be recorded till the end of the surgery, Noninvasive automated arterial blood pressure, heart rate measurements and saturation will be recorded before the spinal anesthesia (baseline), vital data will be monitored 3 minutes after the spinal anesthesia, every 5 minutes in the first 15 minutes after spinal anesthesia, and every 15 min thereafter.

* Hypotension defined as a decrease in Blood pressure (20% from the baseline), will be treated with IV boluses of ephedrine 6 mg repeated every 3 min.
* Bradycardia defined as decrease in the heart rate (20% from the baseline) and Will be treated with atropine 1 mg.
* Desaturation defined as decrease in saturation less than 94% and will be managed by oxygen mask .

C. Postoperative settings:

Monitoring vitals for 12 hours postoperatively for any possible complications every 10 minutes in the PACU and every 30 mins after discharge to the ward unit.

Measurements:

1. Mean arterial Blood pressure (Hypotension defined as decrease in blood pressure 20% from the baseline) will be managed with 6 mg bolus of ephidrine.
2. Heart rate (Bradycardia defined as decrease in heart rate 20% from the baseline ) will be managed with atropine 1mg .
3. Oxygen saturation (Desaturation defined as decrease in saturation below 94%) will be managed with oxygen mask.
4. Incidence complications e.g

   * Nausea and vomiting ( can be managed using metoclopramide).
   * Hypotension ( 6 mg bolus ephedrine will be given).
   * shivering (pethidine 25 mg can be given also dexamethasone 8 mg has an effect in reducing the post spinal shivering)
   * Post dural puncture headache (will be managed by bed rest, IV hydration, caffeine supplementation and analgesics.
   * Spinal hematoma ( will be managed by immediate surgical drainage, vitamin k1 2.5- 10mg and fresh frozen plasma .
   * Total spinal (will be managed by oxygen delivery and intubation).

Statistical Analysis:

● Statistical Package: All data will be analyzed statistically. All data will be included in the SPSS software version 21. The appropriate statistical method will be used for analysis. Descriptive statistics such as mean, standard deviation and percentages will be used. Comparison of categorical data will be done using Chi-square test and for continuous data; unpaired "t" test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Either sex
* 80 to 89 years of age
* undergoing hip surgery

Exclusion Criteria:

* Patient refusal of procedure or participation in the study.

  * Cardiac patients diagnosed with sever Aortic stenosis defined by echo as AVA (aortic valve area) < 1cm and MPG (mean pressure gradient ) >40mmHg.
  * Patients with hemodynamic instability.
  * Preexisting infection at the block site.
  * Allergy to local anesthetics.
  * Psychiatric illness.
  * Increased intracranial tension.
  * Patients with coagulopathy problems.

Ages: 80 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | Intraoperative and up to 12 hours postoperative
  to compare the The incidence of hypotension (defined as decrease in blood pressure 20% from the base line) in continuous spinal anesthesia CSA versus single dose spinal anesthesia in octogenarians undergoing hip surgery

SECONDARY OUTCOMES:
Total use of vasopressor | Intraoperative
  to determine the total use of vasopressor (Ephedrine) in each group
Spinal anesthesia complications | Intraoperative and up to 12 hours postoperative
  the incidence of spinal complications as nausea, vomiting and post dural puncture headache

CONTACTS AND LOCATIONS:
Overall Officials: Hany M. Elzahaby, M.D., Study Director — AinShams University
Locations (1):
- AinShams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol

REFERENCES:
- [Background] Favarel-Garrigues JF, Sztark F, Petitjean ME, Thicoipe M, Lassie P, Dabadie P. Hemodynamic effects of spinal anesthesia in the elderly: single dose versus titration through a catheter. Anesth Analg. 1996 Feb;82(2):312-6. doi: 10.1097/00000539-199602000-00017. PMID 8561333
- [Background] De Andres JA, Febre E, Bellver J, Bolinches R. Continuous spinal anaesthesia versus single dosing. A comparative study. Eur J Anaesthesiol. 1995 Mar;12(2):135-40. PMID 7781632